CLINICAL TRIAL: NCT06782490
Title: A Phase 2, Randomized, Double-Blind, Four-Arm, Placebo-Controlled, Multicenter Study Assessing the Efficacy, Safety and Tolerability of Three Doses of Orally Administered BMS-986368, a FAAH/MAGL Inhibitor, for the Treatment of Spasticity in Participants With Multiple Sclerosis (BALANCE-MSS-1)
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of BMS-986368 in Participants With Multiple Sclerosis Spasticity
Acronym: MSS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM045-1018
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis Spasticity
Keywords: Spasticity; Multiple Sclerosis; BMS-986368
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Administration of BMS-986368 Dose A (Experimental)
  Interventions: Drug: BMS-986368
- Administration of BMS-986368 Dose B (Experimental)
  Interventions: Drug: BMS-986368
- Administration of BMS-986368 Dose C (Experimental)
  Interventions: Drug: BMS-986368
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-986368 — Specified dose on specified days
  Arms: Administration of BMS-986368 Dose A; Administration of BMS-986368 Dose B; Administration of BMS-986368 Dose C
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of BMS-986368 in participants with Multiple Sclerosis Spasticity

ELIGIBILITY:
Inclusion Criteria

* Participants must have a multiple sclerosis (MS) diagnosis.
* Participants must have a history of spasticity due to MS for at least 6 months prior to Visit 1.
* Participants must have a Modified Ashworth Scale (mAS) score ≥2 in each of 2 muscle groups (at least one muscle group in the leg, excluding ankle plantar flexors) at Visit 1.
* Participants must have an Expanded Disability Status Scale (EDSS) score 3.0-6.5 at Visit 1.

Exclusion Criteria

* Participants must not have any concomitant disease or disorder that has symptoms of spasticity or that may influence the participant's level of spasticity.
* Participants must not have an acute MS exacerbation/relapse requiring treatment or alteration in disease modifying drug dose within 3 months of Visit 1 or Visit 2.
* Participants must not have a history of any substance abuse disorder as defined in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Diagnostic Criteria for Drug and Alcohol Abuse.
* Participants must not be currently taking a medication for spasticity that cannot be discontinued and washed out by Visit 2.
* Participants must not have used FAAH/MAGL inhibitor medication or any cannabinoid-related products (including cannabis, cannabidiol (CBD), or tetrahydrocannabinol (THC)) within 30 days prior to Visit 1.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Total Numeric-transformed Modified Ashworth Scale-Most Affected Lower Limb (TNmAS-MALL) score | At week 6

SECONDARY OUTCOMES:
Change from baseline on the Numeric Rating Scale Spasticity (NRS-S) score | At week 6
Change from baseline on the MS Spasticity Scale (MSSS-88) total scores | At week 6
Change from baseline on the Timed 25-Foot Walk (T25FW) score | At week 6
Change from baseline on the Clinical Global Impression of Severity (CGI-S) score | At week 6
Plasma concentrations of BMS-986368 at selected pre- and post-dose time points | Up to week 6
Number of participants with Treatment-Emergent Adverse Events (TEAEs) | Up to week 16
Serious adverse events (SAEs) | Up to week 16
Adverse events (AEs) leading to treatment discontinuation | Up to week 16
AEs leading to death | Up to week 16
AEs leading to clinically significant lab abnormalities | Up to week 16
Number of participants with suicidal ideation and behavior during BMS-986368 administration as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to week 16
Number of participants with withdrawal symptoms following BMS-986368 administration as assessed by the Cannabis Withdrawal Scale (CWS) | Up to week 15

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (54):
- United States (14):
  - Local Institution - 0033, Birmingham, Alabama
  - Perseverance Research Center,LLC, Scottsdale, Arizona
  - Local Institution - 0017, Aurora, Colorado
  - Local Institution - 0068, Naples, Florida
  - USF Health, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Neurology Center of New England, Foxborough, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Local Institution - 0039, Columbus, Ohio
  - Local Institution - 0069, Columbus, Ohio
  - Local Institution - 0067, Philadelphia, Pennsylvania
  - Hope Neurology, Knoxville, Tennessee
  - EvergreenHealth Medical Center, Kirkland, Washington
- Australia (7):
  - John Hunter Hospital, Newcastle, New South Wales
  - University of Sydney - Brain and Mind Research Institute (BMRI), Sydney, New South Wales
  - Centre for Neuroscience Innovation, Kent Town, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Perron Institute, Nedlands, Western Australia
- Canada (6):
  - Local Institution - 0013, Edmonton, Alberta
  - Local Institution - 0024, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Local Institution - 0028, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Lévis, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Czechia (7):
  - Fakultni Nemocnice u sv. Anny v Brne, Brno, Brno-město
  - Local Institution - 0010, Hradec Králové, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague, Praha 2
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Local Institution - 0011, Prague, Praha 5
  - Local Institution - 0053, Pardubice
  - Local Institution - 0009, Teplice, Ústecký kraj
- Germany (9):
  - Klinikum Würzburg Mitte, Würzburg, Bavaria
  - Neurologischen Gemeinschaftspraxis Kassel und Vellmar, Kassel, Hesse
  - St. Josef und St. Elisabeth Hospital gGmbH, Bochum, North Rhine-Westphalia
  - Local Institution - 0060, Münster, North Rhine-Westphalia
  - Local Institution - 0031, Meisenheim, Rhineland-Palatinate
  - Universitätsklinikum Jena, Jena, Thuringia
  - Neurozentrum Bielefeld, Bielefeld
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Local Institution - 0020, Essen
- Poland (10):
  - Centrum Medyczne NEUROMED, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0044, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska Jedynak, Oświęcim, Lesser Poland Voivodeship
  - Local Institution - 0070, Lódz, Lódzkie
  - Centrum Medyczne NeuroProtect, Warsaw, Masovian Voivodeship
  - Local Institution - 0061, Gdansk
  - M.A. - LEK A.M. Maciejowscy S.C., Centrum Terapii SM, Katowice
  - Local Institution - 0051, Słomniki
- Puerto Rico Multiple Sclerosis Center, Caguas, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06782490.html